CLINICAL TRIAL: NCT03524742
Title: Effects of an Avocado Based meDiterranean Diet on Serum Lipids for Secondary Prevention After Ischemic StrokE Trial (ADD-SPISE). Study Protocol.
Brief Title: Effects of an Avocado Based meDiterranean Diet on Serum Lipids for Secondary Prevention After Ischemic StrokE Trial. Study Protocol.
Acronym: ADD-SPISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Alemana de Santiago (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Veronica Olavarria, Principal Investigator, Clinica Alemana de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ADD-SPISE trial
Record Dates: First submitted 2018-04-15; First posted 2018-05-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: Diet; Cholesterol
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Academic, open-label, blinded outcome assessment (PROBE design), clinical trial.
Who Masked: Outcomes Assessor
Masking Description: open-label, blinded outcome assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado-Mediterranean Diet (Experimental): Avocado based Mediterranean diet with intake of ½ portion of a Hass avocado per day, during 3 months.
  Interventions: Other: Avocado-Mediterranean Diet
- Control-Group Diet (Active Comparator): Control-Group Diet consists of a low fat-high complex carbohydrate diet, during 3 months.
  Interventions: Other: Control-Group Diet

INTERVENTIONS:
Other: Avocado-Mediterranean Diet — Mediterranean diet including 1/2 portion of Hass avocado per day, considering a minimum 35% of calories as fat (22% MUFA fat, 6% PUFA fat, and ±10% saturated fat), 15% proteins, and a maximum of 50% carbohydrates.
  Arms: Avocado-Mediterranean Diet
Other: Control-Group Diet — A low fat-high complex carbohydrate diet, during 3 months.
  Arms: Control-Group Diet

SUMMARY:
Recent global burden of disease analysis of DALYs, showed that dietary risk have the highest DALYs in ischemic stroke among behavioral risk factors. The MediDiet is associated with a decreased risk of total mortality as well as stroke incidence and mortality. Although not part of the classical Mediterranean diet they are another nutrient-dense source of MUFA, rich in vitamins, minerals, fiber, phytosterols and polyphenols extensively consumed in the Americas. Avocado-substituted diets significantly decrease cholesterol levels in diabetic and obese patients. Secondary stroke prevention studies with diet as an intervention are lacking and there is little information of what patients eat before or after an ischemic stroke. Lowering Low Density Cholesterol (LDL-C) levels decreases stroke recurrence. The aim is to determine the effect of a Mediterranean style diet based on Avocados on lipid profile particularly LDL-C in patients who have had an ischemic stroke and are at high recurrence risk.Methodology: Academic, open-label, blinded outcome assessment (PROBE design), clinical trial. Participants will be patients with an acute ischemic stroke admitted to Clínica Alemana de Santiago, who fulfills the eligibility criteria. Eligible patients will be randomly assigned to either diet intervention in a 1:1 ratio. The interventions will be: A) Avocado based Mediterranean diet with intake of ½ portion of a Hass avocado per day and B) Standard recommendation of low fat-high complex carbohydrate diet recommended by the National Cholesterol Education Program and the American Heart Association. The main efficacy outcome will be the level of plasma LDL-C level at 3 months of the dietary intervention. Secondary outcomes will be changes in: Levels of serum lipid profile, serum inflammation markers, glycemic control, anthropomorphic measures, stroke recurrence, cardiovascular events, adverse events, compliance. A sample size of 100 patients per group (200 in total) was estimated to provide 80% power and 5% level of significance with 10% loss and 5% crossover to detect the same difference in LDL-C after 3 months of intervention in patients with acute stroke. The investigators hypothesize that an Avocado based Mediterranean diet will significantly reduce levels of LDL-cholesterol at 3 months in patients who have suffered a recent acute ischemic stroke compared to the standard diet.

DETAILED DESCRIPTION:
Introduction: Stroke is the second cause of death and the third of years of life lost worldwide. In Chile, stroke is the second cause of death. Ischemic stroke represents roughly 80% of all strokes. The 11 risk factors responsible for 91.8% of the population attributable risk of ischemic stroke are: Age, Blood Pressure ≥140/90mmHg, smoking, waist to hip ratio, Diabetes Mellitus, physical activity, alcohol intake, psychosocial factors, Apo-lipoproteins, Cardiac causes and noteworthy a healthy diet (35.8% of the population attributable risk). Recent global burden of disease analysis of disability adjusted life years (DALYs), showed that dietary risk have the highest DALYs in ischemic stroke among behavioral risk factors. The MediDiet is associated with a decreased risk of total mortality as well as stroke incidence and mortality. Although not part of the classical Mediterranean diet they are another nutrient-dense source of mono unsaturated fatty acids (MUFA), rich in vitamins, minerals, fiber, phytosterols and polyphenols extensively consumed in the Americas. Avocado-substituted diets significantly decrease cholesterol levels in diabetic and obese patients. Secondary stroke prevention studies with diet as an intervention are lacking and there is very little information of what patients eat before or after an ischemic stroke. Recurrent stroke represent 20% of all ischemic strokes at a population level and depending on the etiology, recurrent stroke can occur from 2 to 20% at 3 months of the initial event. Lowering Low Density Cholesterol (LDL-C) levels decreases stroke recurrence.

Goals: The aim is to determine the effect of a Mediterranean style diet based on Avocados as a source of poli unsaturated fatty acids (PUFAs) on lipid profile particularly LDL-C in patients who have had an ischemic stroke and are at high recurrence risk.

Methodology: Academic, open-label, blinded outcome assessment (prospective, randomized, open-blinded end-point [PROBE design]), clinical trial. Participants will be patients with an acute ischemic stroke admitted to Clínica Alemana de Santiago, who fulfills the eligibility criteria. Eligible patients will be randomly assigned to either diet intervention in a 1:1 ratio. The interventions will be: A) Avocado based Mediterranean diet with intake of ½ portion of a Hass avocado per day and B) Standard recommendation of low fat-high complex carbohydrate diet recommended by the National Cholesterol Education Program and the American Heart Association. The main efficacy outcome will be the level of plasma LDL cholesterol level at 3 months of the dietary intervention. Secondary outcomes will be changes in: Levels of serum lipid profile, serum inflammation markers, glycemic control, anthropomorphic measures of the metabolic syndrome, stroke recurrence, cardiovascular events, adverse events, compliance. A sample size of 100 patients per group (200 in total) was estimated to provide 80% power and 5% level of significance with 10% loss and 5% crossover to detect the same difference in LDL-C after 3 months of intervention in patients with acute stroke. The following measurements will be performed at baseline and at 3 months in all patients: Blood pressure, weight, height, waist circumference, cholesterol and triglyceride levels, glucose level, serum insulin level, Apo- lipoproteins A1 and B levels, soluble intercellular adhesion molecule-1, vascular cell adhesion molecule-1, Apo lipoproteins A and B, and interleukin-6 levels; In a random sample of participants (35%), investigators will measure the oleic acid plasma content as a measure of adherence to Avocado intake.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years.
2. A recent ischemic stroke (within the past month).
3. 1 or more of the following cardiovascular risk factor: hypertension, type 2 diabetes mellitus, insulin resistance, dyslipidemia (elevated LDL or total cholesterol), current tobacco use, coronary heart disease, body mass index ≥25, family history of premature CVD.
4. Informed consent provided.

Exclusion Criteria:

1. Comorbidities that would interfere with compliance of the interventions or low likelihood of changing dietary habits (ie, oncological diseases under chemotherapy, institutionalized patients).
2. Known allergy to avocados.
3. Any feeding limitation that could interfere with the dietary intervention such as dysphagia.
4. Mandatory use drugs for other reasons that can change lipid profile (like hormonal therapy, antiretroviral therapy, chronic steroids etc.).
5. The following ischemic stroke possible etiologies without any of the above mentioned cardiovascular risk factors: arterial dissection, thrombophilia, cerebral vasoconstriction reversible syndrome, other infrequent or rare causes such as vasculitis or stroke related to autoimmune diseases.
6. Any concomitant illness with life expectancy of less than 3 months or that would interfere with the outcome assessments and/or follow-up.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol level | 3 months
  Low Density Lipoprotein (LDL) cholesterol level in mg/dL level at 3 months of the dietary intervention.

SECONDARY OUTCOMES:
Levels of total cholesterol | 3 months
  Total cholesterol level in mg/dL at 3 months of dietary intervention
HDL Cholesterol level | 3 months
  High Density Lipoprotein (HDL) cholesterol level in mg/dL level at 3 months of the dietary intervention.
Triglycerides level | 3 months
  Triglycerides level in mg/dL level at 3 months of the dietary intervention.
Systolic blood pressure | 3 months
  Mean systolic blood pressure in mmHg
Waist to hip ratio | 3 months
  Measure of waist diameter in centimeters and hip diameter in centimeters to report waist to hip ratio
Body mass index | 3 months
  Weight in kilograms and height in meters will be combined to report body mass index in kg/m^2
Serious adverse events | 3 months
  Frequency of serious adverse events
Stroke Recurrence | 3 months
  Frequency of stroke recurrence
Frequency of major cardiovascular events | 3 months
  Frequency of major cardiovascular events (composed by acute myocardial infarction, stroke or vascular death).
ICAM serum level | 3 months
  ICAM (intercelular adhesion molecule) in ng/mL
Interleukin-6 serum level | 3 months
  Level of Interleukin-6 in ng/mL
Apolipoproteins levels A and B | 3 months
  Level of Apolipoporoteins A and B in g/L
VCAM serum level | 3 months
  VCAM (vascular cell adhesion molecule) in ng/mL
Determine plasma oleic acid levels in a subgroup | 3 months
  Measurement of plasma oleic acid levels compared to basal in a randomized sample of 35% of group randomized to avocado based mediterranean diet

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Olavarria, MD, Principal Investigator — Clinica Alemana de Santiago
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Olavarria VV, Campodonico PR, Vollrath V, von Geldern P, Velasquez C, Pavez P, Valente B, Donoso P, Ginesta A, Cavada G, Mazzon E, Navia V, Guzman M, Brinck P, Gallardo A, Gonzalez P, Lavados PM. Efficacy of an avocado-based Mediterranean diet on serum lipids for secondary prevention after ischemic stroke: a randomized phase 2 controlled pilot trial. Lipids Health Dis. 2025 Feb 4;24(1):37. doi: 10.1186/s12944-025-02454-4. PMID 39905430